CLINICAL TRIAL: NCT01293292
Title: Teriparatide (Forsteo) Treatment in Postmenopausal Women: Mechanism of Action. A Two-year Open-label Single-arm Study of Teriparatide in Secondary Care
Brief Title: Teriparatide (Forsteo) Treatment in Postmenopausal Women: Mechanism of Action
Acronym: Forsteo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH15466; 2010-021009-19 (EudraCT Number)
Record Dates: First submitted 2011-02-04; First posted 2011-02-10 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Forsteo; Teriparatide
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Teriparatide — Teriparatide (Forsteo) 20 mcg subcutaneous injection once daily. Duration 104 weeks.
  Other Names: Forsteo

SUMMARY:
Previously the approach to treatment of osteoporosis has been to use medications which prevent excessive resorption of bone. More recently medications that build up new bone, i.e. anabolic treatments, have been, and are being, developed. The investigators would like to develop a strategy for evaluating the effectiveness of anabolic therapies by studying a currently available therapy (teriparatide). This strategy could then be used to assess new anabolic treatments as they are developed for use in humans.

The aims of this study are 1) to fully describe the changes in bone turnover in response to teriparatide by biochemical marker type and by time; 2) to fully describe the changes in bone mineral density (BMD) in response to teriparatide by site, bone compartment and time.

If this study is able to identify an early response to treatment, then this will help speed up drug development in this area, by allowing the identification of promising new anabolic drugs and enabling us to understand their mechanism of action. This will benefit the investigators patients as the investigators will have a better understanding of how these drugs work.

ELIGIBILITY:
Inclusion Criteria

Subjects must:

* Have a bone mineral density T-score (at the lumbar spine or total hip) of less than or equal to -2.5
* Be female
* Be at least 5 years post menopausal (more than 5 years since their last menstrual period) but <85 years old.
* Be ambulatory
* Be able and willing to participate in the study and provide written informed consent
* Have a serum 25(OH)2 vitamin D3 >50 nmol/L (after vitamin D3 loading)

Exclusion Criteria

Patients will not be admitted to the study if they exhibit any of the following:

* Evidence of a clinically significant organic disease which could prevent the patient from completing the study
* A body mass index less than 18 or greater than 35
* Abuse of alcohol or use illicit drugs (information obtained from medical history) or who consumed more than 4 servings of any alcoholic beverage one day prior to the visit (i.e., subjects who might be binge drinkers)
* Any history of cancer within the past 5 years excluding skin cancer non melanomas
* Any history of ongoing conditions or diseases known to cause abnormalities of calcium metabolism or skeletal health including Paget's disease of bone
* Chronic renal disease (as defined by an estimated glomerular filtration rate of ≤ 30mL/min)
* Acute or chronic hepatic disease
* Malabsorption syndromes
* Hyperthyroidism as manifested by TSH outside the lower limit of the normal range
* Hyperparathyroidism
* Hypocalcemia or hypercalcemia
* Osteomalacia
* Cushing's syndrome
* Current use of glucocorticoid therapy
* A corrected serum calcium less than 2.2 mmol/L and a PTH above 100 ng/L (that persists after testing and treatment for vitamin D deficiency)
* A history of any known condition that would interfere with the assessment of DXA at either lumbar spine or femoral neck
* Markedly abnormal clinical laboratory parameters that are assessed as clinically significant by the investigator
* Any previous use of bisphosphonate
* Use any of the following medications within 12 months of starting study drug
* Any fluoride with the exception of use for oral hygiene
* Strontium Ranelate
* Other bone agents (e.g. SERM, isoflavones, HRT)
* Participation in another clinical trial involving active therapy 3 months prior to enrolment
* Less than 5 years since menopause
* Bilateral fractures in the measurement regions (hip, tibia and forearm)
* Recent fracture within the last 12 months
* Prior radiation therapy which may involve the skeleton
* Hypersensitivity to teriparatide or any of its excipients
* Unexplained elevations of alkaline phosphatase
* Any known contraindication to the use of teriparatide

Max Age: 84 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Volumetric bone mineral density (BMD) of the lumbar spine (mg hydroxyapatite/cm3) | 0 to 104 weeks
  Change in volumetric BMD of the lumbar spine (vertebrae L1-3) (mg hydroxyapatite/cm3) measured by quantitative computed tomography (QCT) from 0 to 104 weeks treatment.

SECONDARY OUTCOMES:
Lumbar spine, total hip and whole body bone mineral density (g/cm2) | 0 to 104 weeks
  Changes in lumbar spine, total hip and whole body bone mineral density (g/cm2) measured by dual x-ray absorptiometry (DXA) from 0 to 104 weeks.
Biochemical markers of bone turnover | 0 to 104 weeks
  Changes in biochemcial markers of bone turnover (OC, PINP, bone ALP, urinary NTX, serum CTX, sclerostin, DKK-1) from 0 to 104 weeks.
Distal tibia and radius volumetric body bone mineral density (BMD) (mg hydroxyapatite/cm3) | 0 to 104 weeks
  Changes in distal tibia and radius volumetric bone mineral density (mg hydroxyapatite/cm3) measured by High Resolution peripheral Quantitative Computed Tomography (HR-pQCT) from 0 to 104 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Eastell, MD, FRCP, FRCPath, FMedSci, Study Director — University of Sheffield; Jennifer Walsh, PhD MRCP, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust; Eugene McCloskey, MD, FRCPI, Principal Investigator — University of Sheffield; Nicola Peel, DM FRCP, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust; Angela Rogers, BSc (Hons), PhD, MCSP, Principal Investigator — University of Sheffield; Margaret Paggiosi, Bsc (Hons), PhD, MICR, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust; Lang Yang, PhD CSci, Principal Investigator — University of Sheffield; David Hughes, BMedSci MBChB PhD FRCPath, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust; Mark Wilkinson, PhD, FRCS (Tr&Orth), Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Derived] Gossiel F, Scott JR, Paggiosi MA, Naylor KE, McCloskey EV, Peel NFA, Walsh JS, Eastell R. Effect of Teriparatide Treatment on Circulating Periostin and Its Relationship to Regulators of Bone Formation and BMD in Postmenopausal Women With Osteoporosis. J Clin Endocrinol Metab. 2018 Apr 1;103(4):1302-1309. doi: 10.1210/jc.2017-00283. PMID 29365099